CLINICAL TRIAL: NCT07145398
Title: THE EFFECT OF MANDALA PAINTING ON PAIN, STRESS, AND SLEEP QUALITY IN CHILDREN HOSPITALIZED IN THE BURN UNIT: A RANDOMIZED CONTROLLED STUDY
Brief Title: 69 / 5.000 THE EFFECT OF MANDALA PAINTING ON PAIN, STRESS, AND SLEEP QUALITY IN CHILDREN HOSPITALIZED IN THE BURN UNIT: A RANDOMIZED CONTROLLED STUDY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yusuf GÜRGAN, Student, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Van YuzuncuYıl University
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Burns; Pediatric Burn
Keywords: pediatric burn; mandala painting; paın; stress; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design with pretest-posttest experiment and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Coloring (Experimental): Children hospitalized in the burn unit randomized to this group will participate in daily mandala coloring sessions. Each session will last approximately 30 minutes and will be conducted once per day for 7 consecutive days under the supervision of the research team. During these sessions, children will select and color mandala patterns using crayons or colored pencils. Standard burn unit care will also be provided
  Interventions: Behavioral: Mandala Coloring
- Control - Standard Care (Other): Children in the control group will receive only routine burn unit care without any additional interventions. No mandala coloring sessions will be conducted.
  Interventions: Other: Control - Standard Care

INTERVENTIONS:
Behavioral: Mandala Coloring — Children hospitalized in the burn unit will participate in structured mandala coloring sessions. Each session will last approximately 30 minutes and will be conducted once daily for 7 consecutive days. Children will be provided with printed mandala patterns and coloring materials, and the sessions will be supervised by the research team. The purpose of the intervention is to reduce pain and stress levels and improve sleep quality in burn patients.
  Arms: Mandala Coloring
Other: Control - Standard Care — Children in the control group will receive routine burn unit care without any additional interventions. No mandala coloring sessions will be provided.
  Arms: Control - Standard Care

SUMMARY:
The mandala coloring method allows patients to focus their attention on a circle and use colors with repetitive movements. This state of focus and relaxation can have positive effects on anxiety and other negative moods. There are a limited number of studies in the literature on the use of mandala coloring in children. Therefore, the study was designed to investigate the effects of mandala coloring on pain, stress, and sleep quality in children hospitalized in the burn unit.

DETAILED DESCRIPTION:
Skin is the largest organ in the human body and consists of three layers: the epidermis, dermis, and subcutaneous tissue. A burn is tissue damage resulting from exposure of the skin or subcutaneous tissues to factors such as heat, cold, electricity, chemicals, and radioactive rays. According to the World Health Organization (WHO), burns account for an estimated 180,000 deaths each year, with the majority of these burns occurring in low- and middle-income countries. This situation has become a significant global public health problem.

Children, with their growing and developing physiological and anatomical changes, are considered distinct organisms from adults and are significantly affected by burns. Children are at higher risk of burns due to their delicate skin, age-related differences in motor development, and limited life experiences. In 2017, approximately 84,000 children aged 0-14 were hospitalized for burn treatment in the United States. While scald burns are generally more common in young children, flame burns are more common in adolescents.

Burns are a significant medical condition that can have long-term physical and psychological effects in children. Burn injuries can lead to changes such as trauma, pain, stress symptoms, and sleep disturbances. While some burn cases can be treated on an outpatient basis, interventional procedures performed on patients admitted to a burn unit can cause increased pain. The pain felt during these procedures can sometimes be more severe than the pain felt at the time of injury. The anticipation of pain increases the level of pain felt during therapeutic procedures, creating a vicious cycle in which stress and pain amplify each other.

Sleep quality is also significantly affected in burn patients. Factors such as immobilization methods, therapeutic interventions, mechanical ventilation, and medication use can cause sleep disruption. The most common method for pain management is the use of opioid and non-opioid analgesics. However, long-term opioid use can lead to physical and psychological dependence, respiratory depression, and other side effects. Therefore, integrating non-pharmacological methods into treatment is becoming increasingly important.

Art therapy offers an effective non-pharmacological approach to alleviating the effects of traumatic experiences in children. Mandala painting allows patients to focus their attention on a circle and manipulate colors through repetitive movements. This state of focus and relaxation can have positive effects on anxiety and other negative moods. There are limited studies in the literature using mandala painting in children. Therefore, this study was designed to examine the effects of mandala painting on pain, stress, and sleep quality in children hospitalized in a burn unit.

ELIGIBILITY:
Inclusion Criteria:

* Both the parent and the child are willing to participate in the study.
* Child is between 6 and 12 years of age.
* Burn degree is 1st or 2nd degree.
* The child does not have an acute psychiatric diagnosis (e.g., severe anxiety disorder, psychotic conditions).
* The child has basic fine motor skills (e.g., ability to hold a pencil, ability to color).
* The child does not have any chronic illness.
* The child has newly initiated burn treatment.

Exclusion Criteria:

* Parent or child is not willing to participate in the study.
* Burn degree is 3rd or 4th degree.
* The child has any chronic illness.
* The child has a developmental disorder.
* The child has visual perception impairments (e.g., color blindness, severe visual loss).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-01-04 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Baseline (before the intervention) and day 7
  Pain levels will be assessed using the Wong-Baker FACES Pain Rating Scale, which is validated for children. Scores range from 0 (no pain) to 10 (worst pain).
Stress Level | Baseline and day 7
  Stress levels will be measured using the Perceived Stress Scale for Children (ages 7-11). Higher scores indicate greater perceived stress.
Sleep Quality | Baseline and day 7
  Sleep quality will be evaluated using the Children's Sleep Habits Questionnaire. Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with researchers who provide a methodologically sound proposal. Data will be available upon request beginning 6 months after study completion for a period of 3 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available upon request starting 6 months after study completion for a period of 3 years.
Access Criteria: De-identified individual participant data will be available upon request starting 6 months after study completion for a period of 3 years. Access will be granted to qualified researchers who submit a methodologically sound proposal and sign a data sharing agreement. Supporting documents that may be provided include the study protocol, statistical analysis plan, and informed consent form.